CLINICAL TRIAL: NCT06353880
Title: Effects of Different Types of Obesity on Sperm Quality: A Cross-Sectional Study
Brief Title: Obesity With Sperm Quality in Men With Fertility Need
Status: Not yet recruiting | Type: Observational
Sponsor: Yu xiaowei (Other)
Responsible Party: Sponsor-Investigator, Yu xiaowei, Professor, The First Hospital of Jilin University
Organization: The First Hospital of Jilin University (Other)
Other Study IDs: 24K08-001
Record Dates: First submitted 2024-03-31; First posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Sperm Quality; Obesity; Sex Hormones; Visceral Fat
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Normal BMI Group: Participants with a body mass index (BMI) within the normal range, without obesity-related fat accumulation around the testicles.
  Interventions: Other: Participants will be categorized into three groups based on BMI and the presence of pudendal fat deposition.
- Obese without Pudendal Fat Group: Participants with obesity, characterized by excess adiposity, but without significant accumulation of fat around the testicles.
  Interventions: Other: Participants will be categorized into three groups based on BMI and the presence of pudendal fat deposition.
- Obese with Pudendal Fat Group: Participants with obesity and notable accumulation of fat around the testicles (pudendal fat), contributing to the study of its specific impact on sperm quality.
  Interventions: Other: Participants will be categorized into three groups based on BMI and the presence of pudendal fat deposition.

INTERVENTIONS:
Other: Participants will be categorized into three groups based on BMI and the presence of pudendal fat deposition. — Participants will be categorized into three groups based on BMI and the presence of pudendal fat deposition. Sperm quality parameters, including count, motility, and morphology, will be assessed through semen analysis. Additionally, hormonal profiles related to reproductive health will be evaluated.

SUMMARY:
This study aims to investigate the impact of different types of obesity on sperm quality. Participants will be divided into three groups: a normal BMI group, an obese group without pudendal fat wrapping the testicles, and an obese group with pudendal fat wrapping the testicles. Sperm quality parameters will be compared among these groups to assess potential differences associated with different types of obesity.

DETAILED DESCRIPTION:
Background: Obesity is a well-established risk factor for male infertility, yet the mechanisms underlying this association remain incompletely understood. Recent evidence suggests that the distribution of adipose tissue, particularly pudendal fat deposition, may have distinct effects on male reproductive health beyond overall body mass index (BMI). This cross-sectional study aims to elucidate the differential impact of various obesity types on sperm quality, shedding light on potential pathways for intervention and treatment of male infertility.

Objective: The primary objective of this study is to compare sperm quality parameters among three distinct groups: individuals with a normal BMI, obese individuals without pudendal fat deposition around the testicles, and obese individuals with pudendal fat deposition.

Study Design: This study will employ a cross-sectional design to recruit participants from [insert recruitment settings]. Participants will be categorized into three groups based on BMI and the presence of pudendal fat deposition. Sperm quality parameters, including count, motility, and morphology, will be assessed through semen analysis. Additionally, hormonal profiles related to reproductive health will be evaluated.

Inclusion Criteria: Male individuals with fertility needs with BMI within the specified ranges for normal weight and obesity will be eligible for participation. Participants must provide informed consent prior to enrollment.

Exclusion Criteria: Individuals with known medical conditions affecting fertility, such as cryptorchidism or primary testicular failure, will be excluded from the study. Participants currently undergoing treatment for infertility or with a history of recent exposure to factors known to affect sperm quality (e.g., chemotherapy, radiation therapy) will also be excluded.

Outcome Measures: The primary outcome measure will be the comparison of sperm quality parameters (count, motility, morphology) among the three study groups. Secondary outcome measures will include the evaluation of hormonal profiles related to reproductive health, including levels of testosterone, follicle-stimulating hormone (FSH), and luteinizing hormone (LH).

Sample Size: Cross-sectional study ensures a large sample as far as possible, with a minimum of more than 2000 participants.

Statistical Analysis: Descriptive statistics will be used to summarize demographic characteristics and outcome measures of interest. Group comparisons will be performed using appropriate parametric or non-parametric statistical tests, depending on the distribution of the data. Multivariable regression analysis may be employed to adjust for potential confounding variables.

Ethical Considerations: This study will be conducted in accordance with the principles of the Declaration of Helsinki and local regulatory requirements. Institutional Review Board (IRB) approval will be obtained prior to study initiation. Informed consent will be obtained from all participants, and measures will be taken to ensure confidentiality and privacy throughout the study.

Data Collection and Management: Data will be collected using standardized forms and entered into a secure electronic database. Participant identifiers will be anonymized to protect confidentiality. Data quality checks will be performed regularly to ensure accuracy and completeness.

Study Duration: The anticipated study duration is 12 mons. Recruitment will commence upon IRB approval, with data collection expected to be completed by 2024-6.

Funding: None.

Principal Investigator: Xiaowei Yu

Study Identifier: 24K038-001

ELIGIBILITY:
Inclusion Criteria:

* Male individuals with fertility needs
* BMI within the specified ranges for normal weight and obesity will be eligible for participation.
* Participants must provide informed consent prior to enrollment.

Exclusion Criteria:

* Individuals with known medical conditions affecting fertility, such as cryptorchidism or primary testicular failure.
* Participants currently undergoing treatment for infertility or with a history of recent exposure to factors known to affect sperm quality (e.g., chemotherapy, radiation therapy).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Men who with fertility need.
Study Population: This study will employ a cross-sectional design to recruit participants from a single Reproductive Center at the First Hospital of Jilin University. Participants will be categorized into three groups based on BMI and the presence of pudendal fat deposition. Sperm quality parameters, including count, motility, and morphology, will be assessed through semen analysis. Additionally, hormonal profiles related to reproductive health will be evaluated.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Investigation of Testicular Fat-Wrapped Testes Incidence and Associated Risk Factors | This is a cross-sectional observation study, assessments will be conducted at baseline.
  Criteria for BMI Classification: Weight and height will be combined to report BMI in kg/m^2; Participants will be categorized into normal BMI (<25), obese BMI (≥30), and further subgrouped based on the presence or absence of notable accumulation of fat around the testicles.
  Primary Outcome Measure: Incidence of notable accumulation of fat around the testicles in obese men; Exploration of potential risk factors including lifestyle factors (diet, exercise), comorbidities (diabetes, metabolic syndrome), hormonal imbalances, and genetic predispositions.

SECONDARY OUTCOMES:
Comparison of Sperm Quality Across BMI Categories and Testicular Fat-Wrapped Subgroups | This is a cross-sectional observation study, assessments will be conducted at baseline.
  Criteria for Comparison: Sperm quality parameters will be assessed using standardized methods, including sperm count, motility, morphology, and DNA integrity.
  Outcome Measure: Differences in sperm quality between normal BMI participants, obese participants without testicular fat wrapping, and obese participants with testicular fat wrapping.
Comparison of Sex Hormone Levels Across BMI Categories and Testicular Fat-Wrapped Subgroups | This is a cross-sectional observation study, assessments will be conducted at baseline.
  Criteria for Assessment: Serum levels of testosterone, follicle-stimulating hormone (FSH), luteinizing hormone (LH), and estradiol (E2) will be measured.
  Outcome Measure: Variations in sex hormone levels (testosterone, FSH, LH, E2) between normal BMI participants, obese participants without testicular fat wrapping, and obese participants with testicular fat wrapping.

IPD SHARING:
Plan to Share IPD: Undecided
The entirety of the data supporting article is accessible in textual format, figures, tables, and references. Upon request, additional breakdowns of this data will be promptly provided by the corresponding author.